CLINICAL TRIAL: NCT01430195
Title: Proof of Concept Study to Compare Efficacy and Safety of Subcutaneous, Bioresorbable Afamelanotide Implants and Narrow-Band Ultraviolet B (NB-UVB) Light Versus NB-UVB Light Alone in the Treatment of Nonsegmental Vitiligo
Brief Title: Afamelanotide and Narrow-Band Ultraviolet B (NB-UVB) Light in the Treatment of Nonsegmental Vitiligo (NSV)
Acronym: CUV102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUV102; CUV102 (Other: Clinuvel)
Record Dates: First submitted 2011-08-18; First posted 2011-09-08 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Vitiligo
Keywords: vitiligo; depigmentation; phototherapy; non-segmental vitiligo
MeSH Terms: conditions — Vitiligo | interventions — afamelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afamelanotide + NB-UVB: Experimental (Experimental): Subject in this arm will receive both afamelanotide implants (one implant administered every 28 days, 4 implants in total) and NB-UVB light (administered thrice weekly, 72 treatments in total).
  Interventions: Drug: Afamelanotide
- NB-UVB alone: Active Comparator (Active Comparator): Subjects in this arm will receive NB-UVB light only (administered thrice weekly, 72 treatments in total).
  Interventions: Procedure: Narrow-Band UVB Light Treatment

INTERVENTIONS:
Drug: Afamelanotide — NB-UVB phototherapy with or without subcutaneous, bioresorbable Afamelanotide 16 mg implants, contained in a poly(D,L-lactide-co-glycolide) implant core released over 7-10 days following implantation Other Name: CUV1647
  Other Names: CUV1647
  Arms: Afamelanotide + NB-UVB: Experimental
Procedure: Narrow-Band UVB Light Treatment — To be administered 3 times/week for 6 months. 72 treatments in total.
  Other Names: NB-UVB light treatment
  Arms: NB-UVB alone: Active Comparator

SUMMARY:
The purpose of this study is to look at the efficacy of afamelanotide, when combined with narrow-band ultraviolet B (NB-UVB) light, in patients with nonsegmental vitiligo. Afamelanotide is expected to speed up the repigmentation induced by NB-UVB light, leading to reducing frequency and doses of NB-UVB.

DETAILED DESCRIPTION:
Vitiligo is the most common depigmentation disorder. Interventions in the treatment of vitiligo include phototherapy with narrow-band (NB) ultraviolet B (UVB) irradiation (NB-UVB). Further therapeutic approaches are desired and currently being evaluated. The investigational product, afamelanotide, is a synthetic analogue of the human alpha melanocyte stimulating hormone (alpha-MSH). The earliest described function of alpha-MSH is its ability to stimulate melanin synthesis in the skin and therefore stimulate pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with a confirmed diagnosis nonsegmental vitiligo with 15% to 50% of total body surface involvement
* Stable or slowly progressive vitiligo over a 3-month period
* Aged 18 or more
* Fitzpatrick skin types III-VI
* Willing and able to comply with the conditions specified in this protocol and study procedures in the opinion of the Investigator
* Providing written Informed Consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

* Fitzpatrick skin types I-II
* Vitiligo involving the hands and feet only
* Extensive leukotrichia, in the opinion of the Investigator
* Vitiligo of more than 5 years duration
* Previous treatment with NB-UVB within 6 months prior to the Screening Visit
* Patient not responsive to previous NB-UVB treatment, defined as a patient who has undergone at least 30 NB-UVB sessions with no or minimal clinically relevant pigmentary response, in the opinion of the Investigator
* Allergy to afamelanotide or the polymer contained in the implant or to lignocaine/lidocaine or other local anesthetic to be used during the administration of the implant
* Previous treatment with topical immunomodulators (corticosteroids, calcineurin inhibitors) for vitiligo within 4 weeks prior to the Screening Visit
* History of photosensitivity disorders
* Claustrophobia
* History of photosensitive lupus
* Any active and/or unstable autoimmune disease judged to be clinically significant by the Investigator
* History of melanoma or lentigo maligna
* History of dysplastic nevus syndrome
* Any malignant skin lesions
* Any skin disease that may interfere with the study evaluation
* Any evidence of organ dysfunction or deviation from normal in clinical or laboratory determinations judged to be clinically significant by the Investigator
* History of systemic or psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation
* Female who is pregnant (confirmed by positive β-HCG pregnancy test), are lactating
* Female of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device) during the trial and for a period of three months thereafter
* Sexually active man with a partner of child-bearing potential not using barrier contraception during the trial and for a period of three months hereafter
* Participation in a clinical trial for an investigational agent within 30 days prior to the Screening Visit
* Use of any prior and concomitant therapy which may interfere with the objective of the study, including drugs that cause photosensitivity or skin pigmentation within 60 days prior to the Screening Visit
* Subjects assessed as not suitable for the study in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pigmentation of full body, face, trunk and extremities using the VASI and VETF scores | 6 months

SECONDARY OUTCOMES:
Time to onset of repigmentation of full body, face, trunk and extremities | 6 months
Quality of life using the Dermatology Life Quality Index (DLQI) | 6 months
Vitiligo biopsies assessments (optional, selected sites only) | 6 months
Short term safety of both treatments: Routine laboratory assessments - Full body anterior and posterior photography - Vitiligo lesion photography - Examination of the skin and oral mucosa and digital photography - Ophthalmologic examination | 6 months
Maintenance of pigmentation using the VASI and VETF scores | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry Lim, MD, Principal Investigator — Henry Ford Hospital, 3031 W. Grand Blvd., Suite 800, Detroit, MI 48202, USA
Locations (2):
- United States (2):
  - Henry Ford Medical Center, Detroit, Michigan
  - The Mount Sinai School of Medicine, New York, New York

REFERENCES:
- [Derived] Lim HW, Grimes PE, Agbai O, Hamzavi I, Henderson M, Haddican M, Linkner RV, Lebwohl M. Afamelanotide and narrowband UV-B phototherapy for the treatment of vitiligo: a randomized multicenter trial. JAMA Dermatol. 2015 Jan;151(1):42-50. doi: 10.1001/jamadermatol.2014.1875. PMID 25230094